CLINICAL TRIAL: NCT07061132
Title: Leveraging AI-Powered Interview Simulations to Enhance Employability and Reduce Anxiety in Final-Year Nursing and Midwifery Students: A Randomized Controlled Trial
Brief Title: AI-Powered Interview Simulation to Improve Employability and Reduce Anxiety in Nursing and Midwifery Students
Acronym: CARESIM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Seda Sarikose, Asst. prof., Koç University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2025.203.IRB3.080; 2025.203.IRB3.080 (Other: Koç University Ethics Committee)
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Employment Anxiety; Perceived Employability; Educational Technology; Artificial Intelligence (AI); Nursing Education Research; Midwifery Education; Simulation Training
Keywords: ChatGPT; Artificial Intelligence; Job Interview Simulation; Nursing Students; Midwifery Students; Employability; Interview Anxiety; Self-Efficacy; Simulation-Based Learning

STUDY DESIGN:
Intervention Model Description: Interventional Study Model: Parallel Assignment Model Description: Participants will be randomly assigned to one of two parallel groups. The intervention group will receive a ChatGPT-based job interview simulation, while the control group will receive no intervention. Both groups will complete identical pre- and post-intervention assessments.
Who Masked: Participant, Investigator
Masking Description: Group assignment was concealed using a sealed-envelope method. Randomization was conducted by an independent researcher who was not involved in data collection or intervention delivery. Both participants and investigators were unaware of group allocation until the day of implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Based Interview Simulation Group (Experimental): Arm Description:
  Participants in this arm will complete a structured, AI-powered job interview simulation using ChatGPT-4o. The simulation will consist of nine competency-based questions aligned with international nursing and midwifery standards. The interaction will be conducted individually in written format, and the chatbot will provide short, supportive feedback at the end. No text data will be saved. This simulation is designed to enhance participants' employability perception and reduce their interview-related anxiety.
  Interventions: Other: AI-Based Interview Simulation
- No-Intervention Control Group (No Intervention): Participants in this arm will not receive any intervention during the study period. They will complete the same pre-test and post-test assessments as the intervention group but will not participate in the AI-powered interview simulation. After the study concludes, they may optionally be offered access to the simulation for educational purposes, but no data will be collected from that session.

INTERVENTIONS:
Other: AI-Based Interview Simulation — The intervention group participated in a structured, text-based job interview simulation supported by ChatGPT-4o, using nine standardized prompts based on ICN (2008) and ICM (2024) core competencies. Developed by experts in simulation and nursing education, the intervention aimed to enhance self-efficacy and reduce interview-related anxiety. Each session lasted 15-20 minutes and concluded with structured feedback provided by ChatGPT. Participants were also offered an optional preparation guide with 40 reflective questions across themes such as communication, anxiety, and self-awareness. This preparation was not mandatory and not included in the simulation time.
  Arms: AI-Based Interview Simulation Group

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of a ChatGPT-based job interview simulation on the employment perceptions and interview-related anxiety of senior nursing and midwifery students. Transitioning from education to professional practice in healthcare is a critical phase that directly influences employability and career readiness. Particularly for nursing and midwifery students, the ability to navigate job interviews with confidence plays a pivotal role in shaping their future career paths. As such, innovative and digital interventions are needed to better prepare students for this process.

Grounded in Bandura's Social Cognitive Theory and the Technology Acceptance Model (TAM), the study explores how AI-driven simulations affect students' self-efficacy, perceived utility, and usability, and ultimately their career-related outlook. The intervention involves a structured, text-based job interview simulation powered by ChatGPT-4o, during which students respond to a series of nine professionally tailored questions. These questions are aligned with international competency frameworks such as those from ICN (2008) and ICM (2024), focusing on themes like professionalism, teamwork, evidence-based care, communication, and leadership. At the end of the simulation, the chatbot provides brief, constructive feedback to the participant.

A total of 102 final-year students from Koç University and Istanbul University-Cerrahpaşa will be recruited using stratified randomization. Participants will be assigned to either an intervention group, which will complete the ChatGPT simulation, or a control group, which will not receive any interview intervention but will complete the same pre- and post-test questionnaires. Key outcome measures include the Perceived Future Employability Scale (PFE), the Interview Anxiety Scale (MASI-T), and a simulation experience form for the intervention group. Quantitative data will be analyzed using SPSS with appropriate parametric and non-parametric tests based on data distribution, and an intention-to-treat (ITT) approach will be adopted.

To ensure the integrity of the experiment, blinding procedures, strict confidentiality, and group separation protocols will be applied. The simulation will be conducted individually on research-owned devices in private rooms, and no personal or textual data will be saved from the AI interactions. Ethical approval has been obtained from Koç University Social and Behavioral Ethics Committee. Participation is voluntary, informed consent will be collected, and all processes will comply with the Helsinki Declaration and Turkish Personal Data Protection Law.

Ultimately, this study seeks to offer evidence on the pedagogical utility of AI-based simulation tools in preparing healthcare students for employment, while also contributing to the broader field of digital transformation in health education.

DETAILED DESCRIPTION:
This study introduces an innovative AI-based intervention aimed at enhancing employability preparation among senior nursing and midwifery students through a simulated job interview experience. The intervention is structured around a generative artificial intelligence model (ChatGPT-4o), which delivers a dynamic, text-based interaction mimicking realistic interview settings. The chatbot prompts are informed by international professional competency frameworks and were developed with input from nursing educators, digital learning experts, and HR professionals.

The conceptual basis of the study combines Social Cognitive Theory and the Technology Acceptance Model, allowing exploration of how simulated, interactive environments contribute to professional readiness. In particular, the study investigates the influence of self-efficacy beliefs and user perception of AI technology on employment-related attitudes.

To ensure validity and usability, a pilot implementation was conducted prior to full deployment. This included iterative testing of the chatbot dialogue flow, question clarity, and interview timing, with input from students outside the main sample. Minor refinements were applied to optimize realism and reduce cognitive overload during simulation.

The AI interaction does not involve natural language learning or data retention; its sole function is to facilitate reflective engagement in a structured scenario. All responses are deleted after the session to comply with data protection standards. The chatbot-generated feedback is non-evaluative and designed to reinforce confidence.

Quantitative analysis will be supplemented with descriptive insights from a post-simulation feedback form that captures students' subjective experience, perceived preparedness, and usability impressions. This mixed-methods integration supports a comprehensive understanding of the intervention's practical and pedagogical value.

Ultimately, the project aims to contribute to the responsible implementation of AI tools in health professions education, particularly in the context of employability, professional identity formation, and digital literacy.

ELIGIBILITY:
Inclusion Criteria:

Must be 18 years of age or older

Must be a senior-year student enrolled in a nursing or midwifery program

Must voluntarily agree to participate in the study

Must provide written informed consent

Exclusion Criteria:

Unable to participate in the intervention or assessments due to extended absence or medical leave

Fails to complete either the pre-test or post-test assessments

Previous participation in the pilot phase of the study

Prior exposure to the ChatGPT-based interview simulation used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Future Employability Score | From baseline to post-intervention (approximately 2 weeks)
  Assessed using the Perceived Future Employability Scale (PFE). The scale includes 24 items across 6 subdomains and is rated on a 6-point Likert scale. Higher scores indicate more positive perceptions of future employability. Change in total score from pre-test to post-test will be used to assess the intervention's effect.
Change in Interview Anxiety Score | From baseline to post-intervention (approximately 2 weeks)
  Assessed using the Turkish version of the Measure of Anxiety in Selection Interviews (MASI), originally developed by McCarthy and Goffin (2004) and adapted into Turkish by Turgut, Kümbül Güler, and Vural Yüzbaşı (2024). The scale consists of 30 items across four subscales: communication anxiety, social appearance anxiety, performance anxiety, and behavioral anxiety. Each item is rated on a 5-point Likert scale (1-5). Higher scores indicate higher levels of job interview-related anxiety. Change in total score will be analyzed to evaluate the effectiveness of the intervention.

SECONDARY OUTCOMES:
Simulation Experience Evaluation Score | Immediately after the simulation session
  Participants in the intervention group will complete a post-simulation feedback form designed by the researchers. The form includes 8 closed-ended items rated on a 10-point Visual Analog Scale (VAS) and 3 open-ended questions. Dimensions include realism of the simulation, clarity of chatbot prompts, comfort level, perceived usefulness, performance perception, and readiness for real interviews.

CONTACTS AND LOCATIONS:
Overall Officials: SEDA SARIKOSE, Asst. Prof., Principal Investigator — Koc University School of Nursing
Locations (1):
- Koç University School of Nursing, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to outcome measures will be made available to qualified researchers upon reasonable request, following publication of study results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: These documents may be shared upon publication of the study results or upon reasonable request to the corresponding author.
Access Criteria: Qualified researchers may request access to de-identified supporting documents such as the study protocol, statistical analysis plan, and informed consent form. Requests can be made by contacting the principal investigator via institutional email. Documents will be provided for academic or scientific purposes only, and access may be subject to approval by the research ethics committee.